CLINICAL TRIAL: NCT03601104
Title: Effects of Low Intensity, High Intensity Eccentric Resistance Training Associated With Blood Flow Restriction: a Randomized Controlled Trial
Brief Title: Effects of Low Intensity, High Intensity Eccentric Resistance Training Associated With Blood Flow Restriction
Acronym: oclusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Franciele Marques Vanderle, PhD, Paulista University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 680075683140
Record Dates: First submitted 2018-06-21; First posted 2018-07-26 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Exercise
Keywords: Eccentric Training; Resistance Training
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HIET (n = 15) (Active Comparator): High intensity eccentric training: A high intensity (80% isometric peak) eccentric training of the knee extensors in the isokinetic will be performed during 6 weeks, 3 times a week.
  Interventions: Other: High intensity eccentric training
- HIET-BFR (n= 15) (Experimental): High intensity eccentric training with blood flow restriction (BFR): A high intensity eccentric (80% isometric peak) training of the knee extensors in isokinetic will be performed, associated with a pressure cuff placed in the proximal thigh (40% of absolute occlusion pressure) for 6 weeks, 3 times a week.
  Interventions: Other: High intensity eccentric training with BFR
- LIET-BFR (n = 15) (Experimental): Low intensity eccentric training with blood flow restriction (BFR): A low intensity eccentric (40% isometric peak) training of the knee extensors in isokinetic will be performed associated with a pressure cuff placed in the proximal thigh (40% absolute occlusion pressure) for 6 weeks, 3 times a week.
  Interventions: Other: Low intensity eccentric training with BFR
- LIET (n= 15) (Active Comparator): Low intensity eccentric training: A low intensity (40% isometric peak) eccentric training of the knee extensors in the isokinetic will be performed during 6 weeks, 3 times a week.
  Interventions: Other: Low intensity eccentric training

INTERVENTIONS:
Other: High intensity eccentric training — High intensity eccentric training group with 80% of isometric peak torque.
  Arms: HIET (n = 15)
Other: High intensity eccentric training with BFR — Eccentric high intensity training group with 80% of isometric peak torque associated with blood flow restriction (40% of absolute occlusion pressure).
  Arms: HIET-BFR (n= 15)
Other: Low intensity eccentric training with BFR — Low intensity eccentric training group with 40% of isometric peak torque associated with blood flow restriction (40% of absolute occlusion pressure).
  Arms: LIET-BFR (n = 15)
Other: Low intensity eccentric training — Low intensity eccentric training group with 40% of isometric peak torque
  Arms: LIET (n= 15)

SUMMARY:
Introduction: studies on resistance training of low intensity associated with blood flow restriction in recent years, although there are still gaps that can be explored in relation to their physiological phenomena when associated with eccentric training. In this way, from there the exploration becomes relevant the investigation of eccentric training associated to an RFS. Objective: To analyze and compare the effects of a high intensity and low intensity intensive resistance training associated with an RFS (TREAI-RFS and TREBI-RFS) with a high intensity eccentric resistance training without RFS (TREAI) in knee extensors. Method: The study will consist of 45 male participants, allocated from a stratified randomization into three groups: TREAI (n = 15), TREAI-RFS (n = 15) and TREBI-RFS (n = 15). Participants underwent a training program with a minimum of 40% without RFS, 80% with RFS and 40% with CVS of CVIM, 3 times a week, and the outcomes of muscle strength, muscle structure, power test and Endothelial growth will be assessed one week before, the fourth week and one week after the end of the training program. In addition, clinical markers of perception and recovery effort are investigated before and after a session. The graph used is descriptive and descriptive, as it is used as a model of analysis of variance for the analysis of replications without a two-factor scheme, which provides detailed information on how the measures are repeated, neither. A whole statistical analysis can reach the level of significance of 5%.

ELIGIBILITY:
Inclusion Criteria:

* male sex;
* healthy;
* aged between 18 and 35 years

Exclusion Criteria:

* smokers;
* alcoholics;
* use drugs that influenced cardiac autonomic activity;
* cardiovascular, metabolic or endocrine diseases.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-05-12 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in muscle strength torque peaks at dinamometer isokinetic | baseline, fourth week and one week after sixth week
  The isometric, eccentric and concentric torque peaks will be measured with an isokinetic dynamometer in order to evaluate the adaptations of knee extensor force to eccentric training.
Change in muscular structure with ultrasonography | baseline, fourth week and one week after sixth week.
  Ultrasonographic imaging of the dominant lower limb will be captured to determine muscle thickness of the vastus lateralis (VL) and rectus femoris (RF) muscles.
Change in Vascular Endothelial Growth Factor (VEGF) | baseline, fourth week and one week after sixth week.
  For the analysis of the concentration of endothelial growth factor (VEGF) will be collected 10 ml of blood sample. The plasma of this sample will be stored at -80 ° C for further analysis.
Change in muscle power test | baseline, fourth week and one week after sixth week.
  The strength and muscle power tests will be performed on a vertical squat with a guided bar.

SECONDARY OUTCOMES:
Pain threshold | Assessed at baseline, 4th week, and 6th week.
  To assess the pain threshold, the pressure algometer will be applied at five specific locations on the quadriceps.
Analog Visual Scale | Assessed at baseline, 4th week, and 6th week.
  The subjective evaluation of pain will be obtained through the Visual Analogue Scale (EVA), graded from 0 to 10, with zero being the total absence of pain and 10 the maximum level of pain supported by the participant.
Perceived Effort Scale (Borg) | Assessed at baseline, 4th week, and 6th week.
  The degree of subjective exertion reported by the participants in relation to the lower limbs will be analyzed by Borg's scale of perception of effort of 6 to 20 points, 6 being "very easy" and 20 being "exhaustive."
Recovery Perception Scale | Assessed at baseline, 4th week, and 6th week.
  The perception of recovery of the lower limb submitted to the eccentric exercise protocol will be evaluated by means of a 10-point Likert Scale, where 1 indicates "not recovered" and 10 "fully recovered".

CONTACTS AND LOCATIONS:
Overall Officials: Franciele Marques Vanderlei, PhD, Principal Investigator — Universidade Estadual Paulista - FCT / UNESP
Locations (1):
- Franciele Marques Vanderlei, Presidente Prudente, São Paulo, Brazil